CLINICAL TRIAL: NCT02423304
Title: A Serological Evaluation of 77A/G and 11A/12A Associated Gene Polymorphisms of MMP-13 in Periodontitis Affected and Healthy Individuals
Brief Title: Serological Evaluation of 77A/G and 11A/12A Gene of MMP-13 in Periodontitis Affected and Healthy Individuals
Acronym: SEGPPAH
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre (Other)
Collaborators: Research Institute for Genetic and Human Therapy (Other)
Responsible Party: Principal Investigator, J.surya prasanna, dr.M.Divya Aiswairya, Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre
Other Study IDs: Divya Aiswairya thesis
Record Dates: First submitted 2015-04-17; First posted 2015-04-22 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Generalized Adult Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- test: 50 periodontitis patients
  • Patients will be categorized by Periodontal Disease Index (PDI) by P. Ramfjord(1959) blood samples collected from all patients serum separated and evaluated for77A/G AND 11A/12A associated gene polymorphism of Matrix Metallo Proteinase( MMP)-13 in all the patients. studies showing that there is co relation of these genes with increase inflammation.
  Interventions: Genetic: blood samples collected from all patients
- control: 50 periodontally healthy individuals blood samples collected from all patients serum separated and evaluated for77A/G AND 11A/12A associated gene polymorphism of Matrix Metallo Proteinase (MMP)-13 in all the patients
  Interventions: Genetic: blood samples collected from all patients

INTERVENTIONS:
Genetic: blood samples collected from all patients — blood samples collected from brachial pluxes

SUMMARY:
50 periodontitis 50 healthy individuals serological evaluation will done to see association of 77A/G AND 11A/12A gene polymorphisms of MMP-13

DETAILED DESCRIPTION:
* The study will be conducted on 100 individuals
* 50 chronic periodontitis and 50 healthy individuals will be recruited from the Out Patient Department of Periodontics in the study.
* An informed consent will be obtained from patients who wish to participate in the study.
* Patients will be categorized by Periodontal Disease Index (PDI) by P. Ramfjord(1959)
* After clinical examination, blood samples will be collected and assessed for MMP 13 Gene Polymorphisms.
* Subjects will be selected according to the study criteria and divided into two groups (50 each).

  1. Test group
  2. Control group

ELIGIBILITY:
Inclusion Criteria:• Test group

1. Patients with chronic periodontitis classified according to American Academy of Periodontology ( AAP) 1999
2. Subjects aged between 30-55 years

   * Control group Systemically and periodontally healthy individuals of same age group

Exclusion Criteria:

1. Present and past Smokers
2. Presence of any systemic diseases.
3. Oral diseases other than Periodontitis
4. With a previous history of periodontal treatment in the past 6 months and subjects under any medications.
5. Family history of any diagnosed genetic disorders.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * The study will be conducted on 100 individuals
  * 50 chronic periodontitis and 50 healthy individuals will be recruited from the Out Patient Department of Periodontics in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
to evaluate the association of 77A/G AND 11A/12A gene polymorphism of mmp-13 in periodontitis effected and healthy individuals | 6 months
  collect DNA samples from serum and evaluate for gene polymorphism

REFERENCES:
- [Background] Pirhan D, Atilla G, Emingil G, Tervahartiala T, Sorsa T, Berdeli A. MMP-13 promoter polymorphisms in patients with chronic periodontitis: effects on GCF MMP-13 levels and outcome of periodontal therapy. J Clin Periodontol. 2009 Jun;36(6):474-81. doi: 10.1111/j.1600-051X.2009.01399.x. Epub 2009 Apr 22. PMID 19453573
- [Result] Uitto VJ, Airola K, Vaalamo M, Johansson N, Putnins EE, Firth JD, Salonen J, Lopez-Otin C, Saarialho-Kere U, Kahari VM. Collagenase-3 (matrix metalloproteinase-13) expression is induced in oral mucosal epithelium during chronic inflammation. Am J Pathol. 1998 Jun;152(6):1489-99. PMID 9626053
- [Result] Kiili M, Cox SW, Chen HY, Wahlgren J, Maisi P, Eley BM, Salo T, Sorsa T. Collagenase-2 (MMP-8) and collagenase-3 (MMP-13) in adult periodontitis: molecular forms and levels in gingival crevicular fluid and immunolocalisation in gingival tissue. J Clin Periodontol. 2002 Mar;29(3):224-32. doi: 10.1034/j.1600-051x.2002.290308.x. PMID 11940142
- [Result] Hernandez Rios M, Sorsa T, Obregon F, Tervahartiala T, Valenzuela MA, Pozo P, Dutzan N, Lesaffre E, Molas M, Gamonal J. Proteolytic roles of matrix metalloproteinase (MMP)-13 during progression of chronic periodontitis: initial evidence for MMP-13/MMP-9 activation cascade. J Clin Periodontol. 2009 Dec;36(12):1011-7. doi: 10.1111/j.1600-051X.2009.01488.x. PMID 19929954